CLINICAL TRIAL: NCT06583564
Title: A Single Center Randomized Controlled Study of the Prognosis After Indocyanine Green Fluorescence-guided Radical Surgery in Colorectal Cancer Patients of Stage III
Brief Title: The Prognosis Effect of Indocyanine Green (ICG) Fluorescence Guided Surgery on Disease-free Survival (DFS) of Stage III Colorectal Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Tong Ren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-038-01
Record Dates: First submitted 2024-08-28; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer Stage III
Keywords: Colorectal cancer; Indocyanine green; prognosis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICG group (Experimental): Approximately 0.3 ml of ICG dissolved in 2.5 mg/ml of sterile water was injected submucosally by the endoscopic doctors through colonoscopy at two points around the tumor.All patients underwent standard complete mesocolic excision (CME) or total mesorectal excision (TME) with curable purpose using ICG lymphangiography procedure
  Interventions: Procedure: ICG lymphangiography procedure
- Non-ICG group (No Intervention): All patients underwent standard complete mesocolic excision (CME) or total mesorectal excision (TME) with curable purpose.

INTERVENTIONS:
Procedure: ICG lymphangiography procedure — All patients underwent standard complete mesocolic excision (CME) or total mesorectal excision (TME) with curable purpose using ICG lymphangiography procedure
  Arms: ICG group

SUMMARY:
Previous studies of Indocyanine green (ICG) in colorectal surgery have focused on lymphatic mapping, lymph node detection, and the number of harvested lymph nodes. However, relatively few studies have evaluated the outcomes of this imaging technology, especially the prognosis following of colorectal cancer resection. The present study assessed the prognosis of stage III colorectal cancer patients following ICG fluorescence-guided surgery as compared to conventional surgery without the use of ICG Fluorescence imaging

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years,
* confirmed diagnosis of primary CRC,
* preoperative tumor stage of cT1 to cT4, N+, M0 as determined by contrast-enhanced computed tomography (CT),
* no distant metastasis, and
* American Society of Anesthesiologists(ASA)Physical Status Classification score of 1, 2, or 3

Exclusion Criteria:

* history of previous colorectal surgery, emergent surgery, or palliative resection;
* pregnancy or breastfeeding;
* allergy or history of an adverse reaction to ICG
* severe mental disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-09-27 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) rate | From radical surgery to the end of follow-up ,up to 36 months
  the rate of of no recurrence or metastasis after 3 years from radical surgery

SECONDARY OUTCOMES:
the number of harvested lymph nodes | From radical surgery to the end of perioperative period at 1 month
  the number of harvested lymph nodes of radical surgery
Postoperative complications | From radical surgery to the end of perioperative period at 1 month
  Postoperative complications ICG-related complications, surgery-related complications, and systemic complications. Postoperative complications were graded according to the Clavien-Dindo system
Overall survival rate | From radical surgery to the end of follow-up ,up to 36 months
  the rate of 3 years overall survival after radical surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tongren Hospital, Changning, Shanghai Municipality, China